CLINICAL TRIAL: NCT03524287
Title: Clinical Efficacy of Robotic Total Gastrectomy With D2 Lymph Node Dissection for Locally Advanced Proximal Gastric Cancer：A Prospective Trial
Brief Title: Robotic Total Gastrectomy for Locally Advanced Proximal Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director, Head of gastric surgery, Principal Investigator, Clinical Professor, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-014
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; Robotic Surgery; Spleen-Preserving; No.10 Lymph Node Dissection
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No.10 lymph node dissections (Experimental): Patients with locally advanced upper third gastric carcinoma will performed robotic assisted spleen-preserving No.10 lymph node dissections. After the surgery the patients will be treated with oxaliplatin or platinum-based chemotherapy.
  Interventions: Procedure: Robotic Assisted No.10 Lymph Node Dissections

INTERVENTIONS:
Procedure: Robotic Assisted No.10 Lymph Node Dissections — After exclusion of T4b, bulky lymph nodes, or distant metastasis case et al. Robotic assisted spleen-preserving No.10 lymph node dissections will be performed with curative treated intent in patients with locally advanced upper third gastric adenocarcinoma

SUMMARY:
The purpose of this study is to explore the clinical Efficacy of robotic assisted spleen-preserving No. 10 lymph node dissection for patients with locally advanced upper third gastric adenocarcinoma（cT2-4a, N-/+, M0）.

DETAILED DESCRIPTION:
The incidence of No. 10 lymph node metastasis is high in advanced proximal gastric cancer, reported to range from 9.8%-20.9%, and the presence of No. 10 lymph node metastasis is closely related to survival. Therefore, in East Asia, D2 lymph node dissection of potentially curable locally advanced upper third gastric cancer including No. 10 lymph node is the standard surgical treatment.

Robotic surgery has been developed with the aim of improving surgical quality and overcoming the limitations of conventional laparoscopy in the performance of complex mini-invasive procedures. However, it remains a controversial international issue if it is safe and feasible to conduct robotic assisted spleen-preserving No. 10 lymph node dissection for advanced upper third gastric cancer. There is no prospective study to identify the results.

The study is through a prospective, open, single-arm study,to explore the clinical outcomes of the robotic assisted spleen-preserving No. 10 lymph node dissection in the treatment of locally advanced gastric adenocarcinoma （cT2-4a, N-/+, M0）.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 75 years old
* Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
* Locally advanced tumor in the upper third or middle third of stomach without invading the greater curvature (cT2-4a, N-/+, M0 at preoperative evaluation according to the AJCC (American Joint Committee on Cancer) Cancer Staging Manual Seventh Edition)
* No distant metastasis, no direct invasion of pancreas, spleen or other organs nearby in the preoperative examinations
* Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
* ASA (American Society of Anesthesiology) class I to III
* Written informed consent

Exclusion Criteria:

* Pregnant and lactating women
* Suffering from severe mental disorder
* History of previous upper abdominal surgery (except for laparoscopic cholecystectomy)
* History of previous gastric surgery (including ESD/EMR (Endoscopic Submucosal --Dissection/Endoscopic Mucosal Resection )for gastric cancer)
* Enlarged or bulky regional lymph node （diameter over 3cm）supported by preoperative imaging including enlarged or bulky No.10 lymph node
* History of other malignant disease within the past 5 years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within the past 6 months
* History of cerebrovascular accident within the past 6 months
* History of continuous systematic administration of corticosteroids within 1 month
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
* FEV1<50% of the predicted values
* Splenectomy must be performed due to the obvious tumor invasion in spleen or spleen blood vessels.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
overall postoperative morbidity rates | 30 days
  Refers to the incidence of early postoperative complications. The early postoperative complication are defined as the event observed within 30 days after surgery

SECONDARY OUTCOMES:
Numbers of No.10 lymph node dissection | 9 days
  Numbers of dissected No.10 lymph nodes
Rates of positive No.10 lymph node | 9 days
  The Rates of positive No.10 lymph node are defined as the incidence of positive No.10 lymph node (divide number of positive No.10 lymph nodes by number of total No.10 lymph nodes)
3-year overall survival rate | 36 months
  3-year overall survival rate
3-year disease free survival rate | 36 months
  3-year disease free survival rate
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type
Rates of splenectomy | 1 days
  The Rates of splenectomy are defined as the incidence of splenectomy within operation.
Intraoperative morbidity rates | 1 days
  The intraoperative postoperative morbidity rates are defined as the rates of event observed within operation.
Time to first ambulation | 30 days
  Time to first ambulation in hours is used to assess the postoperative recovery course.
Time to first flatus | 30 days
  Time to first flatus in days is used to assess the postoperative recovery course.
Time to first liquid diet | 30 days
  Time to first liquid diet in days is used to assess the postoperative recovery course.
Time to first soft diet | 30 days
  Time to first soft diet in days is used to assess the postoperative recovery course.
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
The variation of weight | 3, 6, 9 and 12 months
  The variation of weight on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status and quality of life.
The variation of album | 3, 6, 9 and 12 months
  The variation of album in gram/liter on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status and quality of life.
The variation of white blood cell count | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of C-reactive protein | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of C-reactive protein IN milligram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
Technical performance | 1 days
  Technical performance were assessed by the Objective Structured Assessments of Technical Skills (OSATS) and the Generic Error Rating Tool.
The Surgery Task Load Index (SURG-TLX) | 1 days
  Surgeons were required to complete one modified SURG-TLX questionnaire for each procedure.
Lymph node noncompliance rate | 1 days
  Lymph node noncompliance was defined as the absence of lymph nodes that should have been excised from more than 1 lymph node station. Major lymph node noncompliance was defined as more than 2 intended lymph node stations that were not removed.

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhong Q, Zhang ZQ, Yan YQ, Li YF, He QC, Zheng CH, Chen QY, Huang CM. [Long-term oncological safety of robotic total gastrectomy for locally advanced proximal gastric cancer: a 5-year noninferiority comparison based on the FUGES-014 study]. Zhonghua Wei Chang Wai Ke Za Zhi. 2025 Aug 25;28(8):886-894. doi: 10.3760/cma.j.cn441530-20250610-00218. Chinese. PMID 40850834